CLINICAL TRIAL: NCT04298749
Title: A Randomized, Double Blind, Placebo-controlled, Dose-escalation Phase I Study to Investigate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of GX-P1 After Single IV Infusion in Healthy Male Volunteers
Brief Title: Safety and Tolerability of GX-P1 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GX-P1-001
Record Dates: First submitted 2020-02-28; First posted 2020-03-06 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GX-P1 dose level 1 (Experimental): GX-P1 dose level 1
  Interventions: Drug: GX-P1 or Placebo (dose level 1)
- GX-P1 dose level 2 (Experimental): GX-P1 dose level 2
  Interventions: Drug: GX-P1 or Placebo (dose level 2)
- GX-P1 dose level 3 (Experimental): GX-P1 dose level 3
  Interventions: Drug: GX-P1 or Placebo (dose level 3)

INTERVENTIONS:
Drug: GX-P1 or Placebo (dose level 1) — GX-P1 dose level 1 or placebo
  Arms: GX-P1 dose level 1
Drug: GX-P1 or Placebo (dose level 2) — GX-P1 dose level 2 or placebo
  Arms: GX-P1 dose level 2
Drug: GX-P1 or Placebo (dose level 3) — GX-P1 dose level 3 or placebo
  Arms: GX-P1 dose level 3

SUMMARY:
This study is a single-center, double-blind, placebo-controlled, phase I study with healthy male volunteers receiving ascending single dose of GX-P1

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and complying with the requirements of the study and have voluntarily signed the informed consent form (ICF)
2. Healthy male volunteers aged 19-45 years within screening periods
3. Body weight of 50-90 kg, and body mass index (BMI) of 18.0-30.0 kg/m2
4. Healthy subjects as determined by medical history, physical examination vital signs, ECG and clinical laboratory testing

Exclusion Criteria:

1. Any clinical significant pancreatic, hepatic, renal, gastrointestinal, cardiovascular, respiratory, hematological, central nervous system disease or other significant diseases which might influence either the safety of the subject or the absorption, metabolism or excretion of the active agent under investigation
2. History of or current disease evidence including malignant tumor
3. History of allergy/hypersensitivity or ongoing allergy/hypersensitivity to any drug
4. Have participated in another clinical trial with investigational drug within 180 days prior to screening period
5. Positive for HCV antibody, HBsAg, or HIV antibody at screening period
6. Other clinically significant abnormalities which make subject unsuitable for inclusion this study judged by investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by AEs | up to 8 weeks
  Safety and tolerability will be assessed by monitoring AEs and performing physical/clinical examinations

SECONDARY OUTCOMES:
Cmax, Maximum observed concentration | up to 4 weeks
  Maximum observed concentration
Tmax, Time to maximum observed concentration | up to 4 weeks
  Time to maximum observed concentration
T1/2, Elimination half life of GX-P1 | up to 4 weeks
  Elimination half life of GX-P1
AUC(0-inf), Area under the concentration-time curve from time zero extrapolated to infinite time | up to 4 weeks
  Area under the concentration-time curve from time zero extrapolated to infinite time
Change in number of T cells | up to 4 weeks
  Change of T cell subsets
Incidence of Treatment Emergent anti-drug antibody(ADA) formation | up to 8 weeks
  Treatment Emergent anti-drug antibody(ADA) formation

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No